CLINICAL TRIAL: NCT04561180
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of EG-009A Compared to Dexamethasone in Patients With Moderate/Severe (Non-intubated, Non-mechanical Ventilation) COVID-19 Pneumonia
Brief Title: Study to Evaluate the Efficacy and Safety of EG-009A Compared to DEX in Patients With COVID-19 Pneumonia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No patients COVID-19 morbidity decreased.
Sponsor: Evergreen Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HPC-EG-009A-2.1
Record Dates: First submitted 2020-09-22; First posted 2020-09-23 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: COVID-19 Pneumonia
Keywords: COVID 19
MeSH Terms: conditions — COVID-19 | interventions — Standard of Care; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1: SOC + DEX + EG-009A placebo (Placebo Comparator): In addition to the standard of care (SOC), patients will receive dexamethasone (DEX) for 10 days and EG-009A placebo for 3 additional weeks.
  Interventions: Drug: EG-009A Placebo; Drug: Standard of Care; Drug: Dexamethasone
- Arm 2: SOC + DEX + Low Dose EG-009A (Experimental): In addition to the standard of care (SOC), patients will receive dexamethasone (DEX) for 10 days and EG-009A Low dose for 3 additional weeks.
  Interventions: Drug: EG-009A; Drug: Standard of Care; Drug: Dexamethasone
- Arm 3: SOC + DEX + High Dose EG-009A (Experimental): In addition to the standard of care (SOC), patients will receive dexamethasone (DEX) for 10 days and EG-009A High dose for 3 additional weeks.
  Interventions: Drug: EG-009A; Drug: Standard of Care; Drug: Dexamethasone

INTERVENTIONS:
Drug: EG-009A — Administered as an Intramuscular injection
  Arms: Arm 2: SOC + DEX + Low Dose EG-009A; Arm 3: SOC + DEX + High Dose EG-009A
Drug: EG-009A Placebo — Administered as an Intramuscular injection
  Arms: Arm 1: SOC + DEX + EG-009A placebo
Drug: Standard of Care — Standard of Care Treatment for COVID-19 Infection
Drug: Dexamethasone — The comparator, Administered as an Intravenous infusion

SUMMARY:
To study signals of efficacy and safety of a currently available dosage form (IM) of EG-009A in reducing the severity of respiratory disease in patients hospitalized with SARS-CoV-2 virus.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent, or with a legal representative who can provide informed consent, or enrolled under International Conference on Harmonization (ICH) E6(R2) 4.8.15 emergency use provisions as deemed necessary by the investigator (age ≥18), or willing and able to provide assent (age ≥12 to <18, where locally and nationally approved) prior to performing study procedures
2. Patient is aged at least 18 years, enrollment of patients < 65 years old will be limited to 20% of the total with the first 50% of enrollment conducted solely among those patients ≥ 55 years old.
3. Patient has SARS-CoV-2 pneumonia from COVID-19 infection of moderate to serious severity (WHO Ordinal Scale for Clinical Improvement score of 4 or 5)
4. Patient has COVID-19 symptoms ≤ 10 days and at least 1 of the following:

   * Radiographic infiltrates by imaging (chest x-ray, CT scan, etc.)
   * O2 saturation (SpO2) ≤ 94% on room air
   * Requiring supplemental O2 (patients on HFNO ≤ 20 L/min with FiO2 < 0.5 are allowed), but not requiring mechanical ventilation.

Note: Patients admitted with immediate need for mechanical ventilation are of a severity too critical for inclusion into this protocol. Patients who are already in the hospital and have been removed from mechanical ventilation are not eligible.

Exclusion Criteria:

1. Patient has SARS-CoV-2 infection of severity ≥ 6 on COVID-19 WHO Ordinal Scale for Clinical Improvement or for those subjects who have a WHO Ordinal Scale for Clinical Improvement score of 5, nasal intermittent positive pressure ventilation (NIPPV) or requiring HFNO > 20 L/min with FiO2 ≥ 0.5 will be exclusionary.
2. Patient is currently receiving extracorporeal membrane oxygenation, nitric oxide therapy, or high-frequency oscillatory ventilation
3. Patient is unlikely to survive for > 24 hours from randomization, in the opinion of the investigator
4. Patient has a history of chronic oxygen use or any pre-existing respiratory condition that requires intermittent or continuous ambulatory oxygen prior to hospitalization
5. Patient has a history of venous thromboembolism, DVT, or pulmonary embolus
6. Has taken other investigational drugs or participated in any clinical study within 30 days or 5 half-lives (if known) of the investigational drug's PK, PD, or biological activity (if known), whichever is longer, prior to the first dose of study drug in this study or is currently participating in another clinical study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-03-04 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
The proportion of patients alive and without respiratory failure | First dose date to 28 days treatment dosing period
  Patients will be assessed for COVID-19 Ordinal Scale for Clinical Improvement scores and respiratory status throughout the study